CLINICAL TRIAL: NCT04346888
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Pharmacodynamic and Pharmacokinetic of HBM9161 (HL161) Subcutaneous Injection in Patients With Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Efficacy, Safety and PD and PK of HBM9161 in MG Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9161.3
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Myasthenia Gravis
Keywords: MG
MeSH Terms: conditions — Myasthenia Gravis | interventions — HBM9161

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: for double-blind period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBM9161 (680mg and 340 mg) (Experimental): Subcutaneous injection; Blinded: HBM9161 680mg; Open-label: HBM9161 340mg;
  Interventions: Drug: HBM9161 Injection (680mg and 340 mg)
- HBM9161 (340 mg) (Experimental): Subcutaneous injection; Blinded: HBM9161 340mg; Open-label: HBM9161 340mg;
  Interventions: Drug: HBM9161 Injection (340 mg)
- Placebo, HBM9161 (340 mg) (Placebo Comparator): Subcutaneous injection; Blinded: Placebo; Open-label: HBM9161 340mg;
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: HBM9161 Injection (680mg and 340 mg) — HBM9161 Injection (680mg and 340mg)
  Arms: HBM9161 (680mg and 340 mg)
Drug: Placebos — Placebo, HBM9161 Injection (340mg)
  Arms: Placebo, HBM9161 (340 mg)
Drug: HBM9161 Injection (340 mg) — HBM9161 Injection (340 mg)
  Arms: HBM9161 (340 mg)

SUMMARY:
Primary Objectives: To investigate the efficacy of HBM9161 in patients with attack of MG in China

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind and placebo-controlled study. The investigational drug is HBM9161 injection, and the indication is MG.

The subjects will be randomized to three dose groups (340mg, 680mg and placebo) for a 6 weeks' double-blind treatment period followed by an open-label extension treatment period. The study will investigate the safety, efficacy and pharmacodynamic and pharmacokinetic of HBM9161 in patients with attack of MG in China.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Male or female ≥ 18 years of age.
3. A female participant is eligible to participate if she is of:

   1. Non-childbearing potential (physically infertile, including women who have been menopausal for 2 years or more);
   2. Childbearing potential, negative serum pregnancy test results at screening visits, and agree to consistently use acceptable and effective contraceptive methods until 14 days after the final visit.
4. A male participant must take effective contraception during this clinical trial or their heterosexual partner must take effective contraception.
5. Meets MGFA myasthenia gravis clinical classification IIa-IVa (includes types IIa, IIb, IIIa, IIIb, and IVa) at the screening visit and at the baseline visit.
6. Screening and baseline MG-ADL score ≥ 6, and < 50% of them is from ocular muscle.
7. Stable background MG treatments at randomization.
8. Positive serologic test for AChR-Ab or MUSK-Ab at the screening visit and at least 1 of the following:

   1. History of abnormal neuromuscular transmission test demonstrated by sign-fiber-electromyography or repetitive nerve stimulation OR
   2. History of positive edrophonium chloride test OR
   3. Participant has demonstrated improvement in MG signs on oral cholinesterase inhibitors as assessed by the treating physician.

Exclusion Criteria:

1. Use of rituximab, belimumab, eculizumab or any monoclonal antibody/Fc-fusion biologic for immunomodulation within 6 months prior to screening.
2. Immunoglobulins given by SC, IV(IVIG), or intramuscular route, or plasmapheresis/plasma exchange (PE) within 4 weeks before screening.
3. Thymectomy performed < 12 months prior to screening.
4. Total IgG level <6g/L (at screening).
5. Participant has any laboratory abnormality (at screening) that, in the opinion of the investigator, is clinically significant, has not resolved at baseline, and could jeopardize or would compromise the participant's ability to participate in this study.
6. Have known autoimmune disease other than MG that would interfere with the course and conduct of the study (such as uncontrolled thyroid disease).
7. Have an active infection, a recent serious infection (i.e., requiring injectable antimicrobial therapy or hospitalization) within the 8 weeks prior to screening.
8. History of or known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or Mycobacterium tuberculosis. Participants must have negative test results for HBV surface antigen, HBV core antibody, HCV antibody, HIV 1 and 2 antibodies and a negative TB test at screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change in the Myasthenia Gravis Activities of Daily Living (MG-ADL) score from baseline to Day 43 | 43 days
  The MG-ADL profile provides an assessment of MG symptom severity and measures 8 items on a 0-3 scale, with 0 being the least severe. The total sum of the 13 items represents the ADL score. The ADL score can range from 0 (least severe) to 24 (most severe)

SECONDARY OUTCOMES:
Change in the Myasthenia Gravis Composite (MGC) score from baseline to Day 43 | 43 days
  The total QMG score is obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity.
Change in the Quantitative Myasthenia Gravis (QMG) score from baseline to Day 43 | 43 days
  The QMG test is a standardized quantitative strength scoring system and measures 13 items on a 0-3 scale, with 0 being the least severe. The total sum of the 13 items represents the QMG score. The QMG score can range from 0 (least severe) to 39 (most severe).
Change in the Myasthenia Gravis Quality of Life 15(MG-QoL15r) score from baseline to Day 43 | 43 days
  The MG-QoL 15r scale is a patient-reported score that assesses the patient's perception of impairment and disability and the degree to which the patient tolerates disease manifestations. Each question was graded on a 3-point scale from 0=normal to 2=severe with a score of 0 to 30; the higher score indicates worse MG disease activity
Proportion of participants with a decrease on the MG-ADL Score by ≥ 2 points from baseline to Day 43 | 43 days
Proportion of participants with an improvement and worse on the MGFA Post-intervention Status (MGFA-PIS) from baseline to Day 43. o Improvement: MGC Score reduce ≥ 3 points o Aggravation: MGC Score increase ≥ 3 points | 43 days
Change in the MG-ADL score from baseline to Day 120 | 120 days
Change in the MGC score from baseline to Day 120 | 120 days
Change in the QMG score from baseline to Day 120 | 120 days
Change in the MG-QoL15r score from baseline to Day 120 | 120 days
Proportion of participants with persistent improvement on the MGC score from baseline to Day 120 | 120 days
  Improvement (decrease) in the MGC score by ≥ 3 points for 6 weeks
Proportion of participants with persistent improvement on the MG-ADL score from baseline to Day 120 | 120 days
  Improvement (decrease) in the MG-ADL Score by ≥ 2 points for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yan C, Duan RS, Yang H, Li HF, Zou Z, Zhang H, Zhou H, Li XL, Zhou H, Jiao L, Chen J, Yin J, Du Q, Lee M, Chen Y, Chen X, Zhao C. Therapeutic Effects of Batoclimab in Chinese Patients with Generalized Myasthenia Gravis: A Double-Blinded, Randomized, Placebo-Controlled Phase II Study. Neurol Ther. 2022 Jun;11(2):815-834. doi: 10.1007/s40120-022-00345-9. Epub 2022 Apr 12. PMID 35412216

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT04346888/Prot_SAP_000.pdf